CLINICAL TRIAL: NCT04638400
Title: Comparison of Effects of Simvastatin Versus Ezetimibe on Intracellular Lipid and Inflammation in Obese Subjects
Brief Title: Anti-inflammatory Effects of Simvastatin
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of recruitment- Fellow responsible for study graduated
Sponsor: paresh Dandona (Other)
Responsible Party: Sponsor-Investigator, paresh Dandona, Distinguished Professor of Medicine, State University of New York at Buffalo
Organization: State University of New York at Buffalo (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00001035
Record Dates: First submitted 2020-10-07; First posted 2020-11-20 (Actual); Results first posted 2024-01-23 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-10

CONDITIONS: Inflammation; Atherosclerosis; Hypercholesterolemia
MeSH Terms: conditions — Inflammation; Atherosclerosis; Hypercholesterolemia | interventions — Simvastatin; Ezetimibe

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Simvastatin (Active Comparator): Obese subjects with elevated cholesterol
  Interventions: Drug: Simvastatin 40mg
- Ezetimibe (Active Comparator): Obese subjects with elevated cholesterol
  Interventions: Drug: Ezetimibe 10mg

INTERVENTIONS:
Drug: Simvastatin 40mg — Simvastatin administered daily for 6 weeks
  Other Names: Simvastatin
  Arms: Simvastatin
Drug: Ezetimibe 10mg — Ezetimibe administered daily for 6 weeks
  Other Names: Zetia
  Arms: Ezetimibe

SUMMARY:
The purpose of this research study is to determine which of the two ingredients of Vytorin (Simvastatin or Ezetimibe) is responsible for the anti-inflammatory effects of Vytorin

DETAILED DESCRIPTION:
Cardiovascular disease is currently the leading cause of death in the developed countries. Atherosclerosis is the most important cause of cardiovascular disease. Statins are known to exert a powerful anti-atherogenic action which is reflected in a marked beneficial effect on the prevention of cardiovascular effects and cardiovascular mortality. They induce a reduction in the progression and an increase in the regression of atherosclerotic lesions. Statins exert powerful effect on lowering LDLc and are also anti-inflammatory due to their ability to lower CRP concentrations. But little is known about their anti-inflammatory effects at a cellular and molecular levels in humans, in vivo.

Vytorin, a preparation containing simvastatin and ezetimibe, has a powerful effect on lowering LDLc concentration through a combination of effects on the absorption of cholesterol from the gut and hepatic cholesterol biosynthesis. In our previous study we have shown that Vytorin exerts a potent anti-inflammatory effect in the obese in the fasting state and following acute inflammatory changes induced by the intake of cream. The IMPROVE-IT trial, which examined the benefits of adding ezetimibe to simvastatin, showed a small additional benefit of ezetimibe (a 6% reduction in cardiovascular events) compared to simvastatin alone. This is marginal when compared to the established cardiovascular benefits of statins.

We, therefore, explore further into the anti-inflammatory actions of the two components of Vytorin by comparing the effects of simvastatin versus ezetimibe on intracellular lipid and inflammation in obese patients to determine which of the two ingredients of Vytorin is responsible for the specific combination of these effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years of age.
2. Obese (BMI ≥30 kg/m2)
3. LDL cholesterol of ≥100 mg/dl
4. Not taking any vitamins or antioxidants

Exclusion Criteria:

1. Currently using anti-hyperlipidemic therapies
2. Triglycerides >500 mg/dl.
3. Myocardial infarction, angioplasty/stent placement or coronary artery bypass surgery in the past 6 months.
4. Patient on chronic use of non-steroidal anti-inflammatory drugs or steroids
5. Hepatic disease
6. Renal impairment.
7. History of drug or alcohol abuse
8. Participation in any other concurrent clinical trial
9. Use of an investigational agent or therapeutic regimen within 30 days of study.
10. Smoker
11. Pregnancy
12. Premenopausal women who are not on birth control pills and have not had a hysterectomy or tubal ligation
13. Anemia with hemoglobin <12 g/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paresh Dandona, MD, PhD, Principal Investigator — Distinguished Professor of Medicine
Locations (1):
- Diabetes and Endocrinology Research Center of WNY, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simvastatin | Ezetimibe
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simvastatin | Ezetimibe | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (4.2) | 53.2 (4.2) | 53.2 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 2 | 1 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10
Change in CD68 mRNA expression [Mean (Standard Deviation); unit: Percent of Change] | 48 (11) | 44.5 (7) | 46 (9)

OUTCOME MEASURES:

1. Primary Outcome: Change in mRNA Expression of CD68 in MNC
Description: Percentage change in mRNA expression of CD68 in MNC following cream challenge at weeks 0 and 6 of treatment with simvastatin or ezetimibe.
  Percent change (using the formula: (x-y)/y*100) is calculated using data collected before (0hr) and after the cream challenge (peak effect) at weeks 0 and 6 of treatment with simvastatin or ezetimibe.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 5 | 5
percentage change
  week 0 | 48 (11) | 44.5 (7)
  week 6 | 38 (9) | 35 (5)

2. Primary Outcome: Change in mRNA Expression of PECAM on MNC
Description: Percentage change in mRNA expression of PECAM on MNC following cream challenge before and after 6 weeks of treatment with simvastatin or ezetimibe. Percent change (using the formula: (x-y)/y*100) was calculated using data collected before (0hr) and after the cream challenge (peak effect) at weeks 0 and 6 of treatment with simvastatin or ezetimibe.
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 5 | 5
percentage change
  week 0 | 38 (8) | 42 (6)
  week 6 | 36 (10) | 38 (8)

3. Secondary Outcome: Change in mRNA Expression of IL-1β in MNC
Description: Percentage change in mRNA expression of IL-1β in MNC following cream challenge calculated from data collected before (at 0 week) and after (at 6 weeks) treatment with simvastatin or ezetimibe
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 5 | 5
percentage of change
  week 0 | 41 (15) | 38 (11)
  week6 | 36 (7) | 40 (12)

4. Secondary Outcome: Change in TNF-a mRNA Expression in MNC
Description: Percentage change in mRNA expression of TNFα in MNC following cream challenge calculated using data collected before and after the cream challenge at weeks 0 and 6 of treatment with simvastatin or ezetimibe
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 5 | 5
percentage of change
  week 0 | 48 (17) | 43 (9)
  week 6 | 41 (13) | 38 (6)

5. Secondary Outcome: Change in mRNA Expression of MMP-9 in MNC
Description: Percentage change in mRNA expression of MMP-9 in MNC calculated from data collected following cream challenge before (0 week) and after (6 weeks) of treatment with simvastatin or ezetimibe
Time Frame: 6 weeks
Measure: Mean (Standard Error); unit: percentage of change
Arm/Group | Simvastatin | Ezetimibe
Number analyzed (Participants) | 5 | 5
percentage of change
  week 0 | 34 (8) | 35 (6)
  week 6 | 28 (12) | 36 (8)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Simvastatin | Ezetimibe
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT04638400/Prot_SAP_002.pdf